CLINICAL TRIAL: NCT02520323
Title: The Lung Microbiome in Sarcoidosis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Eric S. White, MD, Associate Professor, University of Michigan
Other Study IDs: HUM00095799
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Blood Specimen Collection; Bronchoscopy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blood only: 20 sarcoidosis subjects and 20 healthy controls will complete lifestyle questionnaires and have blood drawn for microbiome analyses.
  Interventions: Other: Blood draw; Behavioral: Questionnaires
- Blood and BAL: 10 sarcoidosis subjects, 10 healthy controls, and 10 subjects with non-sarcoid interstitial lung disease will complete lifestyle questionnaires and undergo blood sampling for microbiome analyses as well as bronchoscopy for bronchoalveolar lavage microbiome analyses.
  Interventions: Other: Blood draw; Procedure: Bronchoscopy; Behavioral: Questionnaires

INTERVENTIONS:
Other: Blood draw
Procedure: Bronchoscopy
  Groups: Blood and BAL
Behavioral: Questionnaires

SUMMARY:
The objective of this study is to determine the presence of bacterial species, and the immunologic and molecular mechanisms of granuloma formation that might be involved in the pathogenesis of sarcoidosis. The investigators will collect peripheral blood and bronchoalveolar lavage fluid samples to isolate bacterial DNA and blood monocytes and lymphocytes. Specimens will be obtained from patients with sarcoidosis, with non-sarcoid lung disease, and healthy volunteers to directly compare the bacterial species present and the characteristics of cells thought to be involved in granuloma formation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sarcoidosis (30 subjects) or
* Clinical diagnosis of non-sarcoid interstitial lung disease (10 subjects) or
* Age-matched controls (30 subjects)
* Ability to provide informed consent

Exclusion Criteria:

* Any disease condition (such as anemia, unstable cardiac disease, etc.) that in the opinion of the subject's primary physician would put the patient at risk of harm from having 60 cc of blood drawn or for undergoing bronchoscopy for this study.
* Patients who are undergoing bronchoscopy for presumed infection.
* Pregnant women, women who may be pregnant, and women who are breastfeeding.
* Patients who have undergone lung transplantation.
* Persons who are unable or unwilling to undergo bronchoscopy, including those unable to be accompanied by a designated driver to the procedure.
* Persons who have taken antibiotics in the 90 days prior to consent.
* Known HIV, HCV, alcohol, or other substance abuse history.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Potential subjects will be patients with sarcoidosis (involving any organ system), with non-sarcoid interstitial lung disease, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Microbiome analysis | Baseline
  To assess the microbiome profile in lung lavage fluid and peripheral blood of subjects

SECONDARY OUTCOMES:
Measures of immunologic phenotype | Baseline
  To determine whether the immune cell profile of sarcoidosis patients differs from healthy controls and other interstitial lung disease patients in blood and BAL fluid

CONTACTS AND LOCATIONS:
Overall Officials: Eric S White, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States